CLINICAL TRIAL: NCT04269265
Title: The Effect of Inflammation and Damage to Lymph Node Structures on Durable Protective Immunity Following Yellow Fever Vaccination
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IDIM-2018-27222; U01AI141981 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All Participants (Experimental): In this single-arm study, all participants will receive the intervention
  Interventions: Biological: Yellow Fever Vaccine

INTERVENTIONS:
Biological: Yellow Fever Vaccine — YF-VAX®, Yellow Fever Vaccine, for subcutaneous use
  Other Names: YF-VAX

SUMMARY:
Hypothesis: Infections other than HIV can cause LN inflammation and collagen damage to the fibroblastic reticular cell network (FRCn), which will lead to CD4 T cell depletion and impaired vaccine responses. This protocol will study yellow fever vaccine (YFV) in two cohorts of people, one from Uganda and the other from Minnesota where we collect lymphoid tissues (LT) and peripheral blood monocytes (PBMCs) before and after vaccination using a new technique to catalog infectious burden of the individual, determine the relationship between IA, Infections, and immune response.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the difference between antibody titers in the two study groups and study the relationship between endemic infections, IA, the FRCn, and CD4 and CD8 T cell subsets and the magnitude and durability of neutralizing antibody response to YFV in a cohort shown to have elevated IA, a damaged FRCn, and pan T cell depletion and a cohort that does not. This is a single arm, open-label, two cohort study of healthy adults in Kampala, Uganda and in Minnesota, USA. The cohort in Uganda will be 30 adults (15 men and 15 women) and the cohort in Minnesota will be 16 adults (8 men and 8 women). Everyone will be screened to ensure there are no contraindications to receiving YFV (e.g., immunosuppression) or the planned procedures. The inclusion and exclusion criteria are discussed in detail in the protocol that is included in the appendix. Participants will have an inguinal lymph node and adjacent adipose tissue biopsy and leukapheresis prior to YFV and again 3 weeks after the vaccine administration. The vaccine will be given in the contralateral thigh from the first LN biopsy so that the second biopsy will be from a draining LN. PBMC and plasma as well as urine and stool will be collected at regular intervals over the 18-month follow-up period and leukapheresis will be done again at the month 18 visit.

ELIGIBILITY:
Inclusion Criteria:

* No contraindication to Yellow Fever vaccine (immunosuppressed for any reason or on an immunosuppressive drug where a live virus vaccine is contraindicated).
* If female of childbearing age must agree to contraception for one month following administration of the vaccination.

Exclusion Criteria:

* History of yellow fever or previous vaccination for yellow fever
* Known bleeding disorder
* Prior surgery complicated by clotting abnormality
* Psychiatric or behavioral disorder that, in the opinion of the investigator, will make it difficult for the participant to complete the study
* History of acute hypersensitivity reaction to any component of the vaccine (including gelatin, eggs, egg products, or chicken protein).
* Thymus disorder associated with abnormal immune function
* Immunosuppression from any of the following: HIV infection or AIDS, malignant neoplasms, primary immunodeficiencies, transplantation, transplantation, immunosuppressive or immunomodulatory therapy (corticosteroids, alkylating agents, antimetabolites, TNF inhibitors, IL-1 blocking agents, monoclonal antibodies targeting immune cells), previous radiation therapy.
* Pregnant or breastfeeding at the time of vaccination.
* Planning to conceive within 28 days of enrollment and vaccination with the yellow fever vaccine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- Joint Clinical Research Centre, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 43
Completed | 37
Not Completed | 6
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Overenrolled (sample size reached) | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 3
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Neutralizing Antibody Titer
Description: Peak titer of neutralizing antibody to yellow fever vaccination. Outcome reported as Log YF Antibody titer.
Time Frame: 18 months
Measure: Geometric Mean (95% Confidence Interval); unit: Log YF antibody titer
Arm/Group | All Participants
Number analyzed (Participants) | 37
Log YF antibody titer | 1.37 [1.06 to 1.69]

ADVERSE EVENTS:
Time Frame: Through study completion (up to 18 months).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 24/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=37)
Pain at Incision Site (Nervous system disorders) | 8 (8)
Infection at Incision Site (Infections and infestations) | 7 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (5)
Bruising at Incision Site (Blood and lymphatic system disorders) | 3 (3)
Bruising at Venipuncture Site (Blood and lymphatic system disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04269265/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT04269265/ICF_000.pdf